CLINICAL TRIAL: NCT00402480
Title: Effects of Hydroxyurea on the Prevention of Primary Stroke in Children With Sickle Cell Anemia and Elevated Transcranial Doppler (TCD) Flow Velocity
Brief Title: Hydroxyurea to Prevent Stroke in Children With Sickle Cell Anemia and Elevated TCD Flow Velocity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4744
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2006-11

CONDITIONS: Stroke
Keywords: Sickle Cell Anemia with Elevated TCD flow velocity
MeSH Terms: conditions — Stroke | interventions — Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea

SUMMARY:
The purpose of this study is to assess prospectively the efficacy of hydroxyurea therapy in the setting of cerebrovascular disease, manifest as conditional or abnormal transcranial doppler ultrasonography (TCD) flow velocities, in children with sickle cell anemia (SCA). TCD is used to measure flow velocity in intracranial arteries as a marker of increased stroke risk in children with SCA. The primary objective of this protocol is to determine whether hydroxyurea reduces elevated TCD velocity.

DETAILED DESCRIPTION:
The purpose of this study is to assess prospectively the efficacy of hydroxyurea therapy in the setting of cerebrovascular disease, manifest as conditional or abnormal transcranial doppler ultrasonography (TCD) flow velocities, in children with sickle cell anemia (SCA). TCD is used to measure flow velocity in intracranial arteries as a marker of increased stroke risk in children with SCA. The primary objective of this protocol is to determine whether hydroxyurea reduces elevated TCD velocity.

The STOP (Stroke Prevention in Sickle Cell Anemia) trial, a multicenter, randomized, controlled trial for primary stroke demonstrated that monthly blood transfusions, when compared to observation alone, significantly reduced the risk of primary stroke for children with SCA whose TCD velocity exceeded 200 cm/sec. Despite the STOP trial's clear results, there are unresolved issues regarding TCD and stroke risk in children with SCA. First, the predictive value of an abnormal result is not compelling since less than a third of children with an abnormal TCD velocity and even fewer with conditional results will ever develop a clinical stroke. There is also discordance between TCD and MRI results. Only 40% of children with abnormal TCD velocity will have abnormalities on brain MRI (Wang, et al. J Pediatr Hematol/Oncol 2000;22(4):335-339, Pegelow, et al. Arch Neurol 2001;58:2017-2021). There are also well recognized risks of chronic blood transfusions, including iron overload and alloimmunization, and the necessary duration of transfusion protection for children with abnormal TCD velocity is unknown. Unfortunately, there are currently no therapeutic options besides blood transfusions for patients with SCA and an abnormal TCD velocity.

Erythrocyte transfusions and hydroxyurea have many similar beneficial effects in patients with SCA. Transfusions may prevent primary stroke by lowering the % HbS, by increasing the hematocrit, by improving red cell rheology, by decreasing red cell adhesion, and by lowering TCD velocity. Hydroxyurea leads to many of the same changes, thus in this protocol, we will examine whether hydroxyurea, like transfusions, can lower TCD velocity. In our patients with SCA who have been screened with TCD ultrasonography, we have observed that children who were screened while receiving hydroxyurea had lower TCD velocity measurements than those who were not on hydroxyurea. In a small number of patients with TCD velocity measurements before and after initiation of hydroxyurea for non-neurological reasons, the TCD velocity declined significantly after achieving full dose hydroxyurea therapy. The changes in TCD velocity were correlated with changes in hematocrit since hydroxyurea increases blood counts in patients with SCA. For each % increase in hematocrit, the TCD velocity increased by 6.3 cm/sec. This was similar to an abstract from the STOP trial, in which TCD flow velocity declined by 7.9 cm/sec for each increase in % hematocrit from transfusions.

Based on this preliminary data, we initiated this prospective, single-institution, pilot trial to determine whether hydroxyurea therapy lowers TCD flow velocity in children with sickle cell anemia.

ELIGIBILITY:
Inclusion Criteria:

* Children with Sickle Cell Anemia
* Aged 3 to 18 years
* Confirmed TCD velocity greater than or equal to 140cm/sec
* Negative serum pregnancy test for subjects of childbearing potential
* Decline transfusions (for subjects with TCD velocity greater than or equal to 200 cm/sec)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2003-04; Study Completion 2006-03

PRIMARY OUTCOMES:
Change in TCD flow velocity

SECONDARY OUTCOMES:
Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Zimmerman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States